CLINICAL TRIAL: NCT05886985
Title: A Phase I Open-Label, Dose-Escalation Study to Evaluate Safety, Tolerability, and Efficacy of Allogeneic Placenta-derived Human Mesenchymal Stem Cells for the Treatment of Acute Respiratory Distress Syndrome
Brief Title: Safety, Tolerability, and Efficacy of MatriPlax in Subjects With Acute Respiratory Distress Syndrome
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BioSpring Medical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-01
Record Dates: First submitted 2023-05-24; First posted 2023-06-02 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: MatriPlax
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MatriPlax (Experimental): Each subject will receive 2x10^7, 4x10^7, or 8x10^7 pcMSCs per administration
  Interventions: Drug: MatriPlax

INTERVENTIONS:
Drug: MatriPlax — MatriPlax contains pcMSCs (placenta choriodecidual membrane-derived mesenchymal stem cells) and will be given intravenously on Day 1 and Day 4
  Other Names: Placenta choriodecidual membrane-derived mesenchymal stem cells

SUMMARY:
The goal of this clinical trial is to explore the safety, tolerability, and efficacy in study intervention, MatriPlax, in subjects with Acute Respiratory Distress Syndrome (ARDS). MatriPlax contains placenta choriodecidual membrane-derived Mesenchymal Stem Cells (pcMSCs). Participants will receive two doses of MatriPlax on Day 1 and Day 4 and conduct efficacy and safety evaluations until 12 months after treatment or withdrawal from the study.

DETAILED DESCRIPTION:
This open-label, dose-escalation Phase I study plans to evaluate the safety, tolerability, and efficacy of MatriPlax.

This is a conventional 3+3 dose-escalation study in which subjects with moderate or severe ARDS will receive intravenous MatriPlax infusion.

Participants will be assigned to one of three dose cohorts (low, middle and high doses of MatriPlax), depending on the time of their enrollment. Each participant will receive two doses of MatriPlax on Day 1 and Day 4. Each dose cohort will have three to six subjects enrolled sequentially with at least 1 week in between. All participants will be followed until 12 months after receiving MatriPlax or withdrawal from the study.

A Data Safety and Monitoring Board (DSMB) meeting will be held when all participants of each cohort complete their 28-day of treatment and evaluation period. The DSMB will determine if the study is safe to proceed to the next dose level or it requires to recruit more subjects to the concurrent dose level for safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of moderate or severe ARDS according to the Berlin definition

   * Acute onset of respiratory failure within 1 week of identified insult
   * Respiratory failure associated with known ARDS risk factors and not fully explained by either cardiac failure or fluid overload
   * Radiological abnormalities on chest X-ray or computerized tomography (CT) scan, i.e., bilateral infiltrates that are not fully explained by effusions, lobar/lung collapse, or nodules
   * Hypoxic respiratory failure

     * Moderate ARDS: PaO2/ FiO2 ratio > 100 mmHg (13.3 kPa) to ≤ 200 mmHg (26.6 kPa) with positive end expiratory pressure (PEEP) ≥ 5 cmH2O
     * Severe ARDS: PaO2/ FiO2 ratio ≤ 100 mmHg (13.3 kPa) with PEEP ≥ 5 cmH2O
2. Administration of study drug must be planned to take place within 72 hours since moderate or severe ARDS diagnosis
3. Either gender, 20 ~ 80 years old (inclusive)
4. Dated and signed informed consent
5. A subject has been admitted to an ICU or RCC and is already on or candidates for mechanical ventilation
6. A subject with the primary disease of ARDS caused by documented virus infection (including severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2))
7. With normal vital sign parameters:

   1. Systolic blood pressure ≥ 90 mmHg and ≤ 160 mmHg
   2. Diastolic blood pressure ≥ 50 mmHg and ≤ 95 mmHg
   3. Pulse rate ≥ 60 beats per minute (bpm) and ≤ 100 bpm
   4. Body temperature ≥ 35.5°C and ≤ 37.7°C

Exclusion Criteria:

1. No intent/unwillingness to follow lung-protective ventilation strategy or fluid management manual
2. On extracorporeal membrane oxygenation (ECMO) support
3. Severe chronic respiratory disease with a PaCO2 > 50 mm Hg or with any oxygen support
4. A subject who is extremely unlikely to survive more than 24 hours in the opinion of the investigator
5. World Health Organization (WHO) Class III or IV pulmonary hypertension
6. Clinical evidence of left ventricular failure
7. With acute diseases or serious medical conditions include cardiovascular (such as cardiac arrhythmia, QT prolongation), pulmonary (except ARDS), hepatic, neurologic, metabolic, renal, psychiatric condition, autoimmune disease, medical history, physical findings, or laboratory abnormality that in the investigators' opinion are not in stable condition and participating in the study could adversely affect the safety of the subject
8. Severe liver disease (Childs-Pugh Score > 10)
9. Acute or chronic kidney disease (Stage-3B, 4 or 5 renal impair; estimated glomerular filtration rate (eGFR) ˂ 60 mL/min/1.73 m^2 or dialysis)

   Note: eGFR (mL/min/1.73 m^2) = 186.3 × (serum creatinine in mg/dL)^-1.154 × (age)^-0.203× (0.742 if female) × (1.212 if African American/black)
10. History of pulmonary embolism
11. Previous solid organ transplant
12. With major surgery within 14 days prior to Screening visit Note: Major surgery is defined as an invasive operative procedure where one or more of the following occurred: 1) A body cavity was entered; 2) A mesenchymal barrier was crossed; 3) A fascial plane was opened; 4) An organ was removed; 5) Normal anatomy was operatively altered. All other invasive operative procedures are minor surgeries.
13. Presence of any active malignancy within 2 years prior to Screening visit
14. History of the human immunodeficiency virus (HIV) infection
15. History of severe allergic or anaphylactic reactions
16. Known or suspected hypersensitivity or previous adverse reaction to any ingredients of study product
17. Participation in a clinical trial of an interventional medicinal product within 12 weeks prior to Screening visit
18. With any other uncontrolled illness judged by the principal investigator that entering the trial may be detrimental to the subject
19. Pregnant or lactating or premenopausal with childbearing potential but not taking reliable contraceptive method(s) during the study period. At least one form of birth control must be adopted. Acceptable forms include:

    * Placement of an intrauterine device (IUD) or intrauterine system (IUS).
    * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps)
20. Female subject with childbearing potential who has positive serum or urine pregnancy test at Screening Visit
21. Unable to return for follow-up visits for clinical evaluation or laboratory studies
22. Inappropriate to participate in this clinical study because of psychiatric disorders or any condition as judged by the principal investigator
23. Hypersensitive to penicillin, streptomycin and amphotericin B antibiotics
24. With specific known risk factors for thrombotic events, including obesity (Body mass index (BMI) >35), diabetes mellitus Type I, history of deep vein thrombosis (DVT) or thrombotic episodes, acquired or inherited thrombophilic disorders, hypercoagulable conditions, and other cardiovascular risk factors judged by the investigator
25. Use of estrogens/oral contraceptives within 6 weeks prior to Screening visit
26. Current smoker or has smoked within 3 months prior to Screening visit.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
The incidence of treatment-emergent adverse events (TEAEs) up to 28 days after receiving MatriPlax | Day 1 to Day 29
  TEAEs are adverse events (AE) that occur after the study intervention administration
The incidence of serious adverse events (SAEs) up to 28 days after receiving MatriPlax | Day 1 to Day 29
  SAE is an AE that results in any of the following outcomes: Death; Life-threatening; Requires inpatient hospitalization or prolongation of existing hospitalization; Results in persistent or significant disability/incapacity; Congenital anomaly/birth defect; Based upon appropriate medical judgment, the event may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed above
The incidence of suspected unexpected serious adverse reactions (SUSAR) up to 28 days after receiving MatriPlax | Day 1 to Day 29
  SUSAR is an SAE that is considered related to study intervention and unexpected judged by sponsor and investigator

SECONDARY OUTCOMES:
Changes in PaO2/FiO2 ratio from baseline | Baseline, Day 4, 6, 8, 15, 29
  The PaO2/FiO2 ratio is the ratio of arterial oxygen partial pressure (PaO2) to fractional inspired oxygen (FiO2), which is an indicator of the severity of ARDS.
Changes in Lung injury score (LIS) from baseline | Baseline, Day 8, 29
  The LIS is a standard measure of ARDS, which is composed of four components. Each component has 5 scores (0, 1, 2, 3 and 4-point) and the score of LIS is the average of the four components. A higher LIS indicates more severe lung injury.
Overall survival | Baseline, Day 29, Month 3, 6, 9, 12
  Overall survival is defined as the time from treatment to death.
All-cause mortality rate | Baseline, Day 29, Month 3, 6, 9, 12
  All-cause mortality rate is defined as the rate of deaths from any cause in all participants.
Cumulative ventilator-free hours (VFH) | Day 1 to 29
  Only subjects who wean from the ventilator and have at least 48 consecutive weaning hours
Time to the first weaning from ventilator | Up to 12 months
  Only subjects who wean from the ventilator and have at least 48 consecutive weaning hours
Number of subjects weaned from ventilator | Day 29
  Only subjects who wean from the ventilator and have at least 48 consecutive weaning hours
Intensive Care Unit (ICU) free hours | Day 1 to 29
  Only subjects who are stable for discharge from ICU and have at least 48 consecutive hours of discharge
Time to the first ICU discharge | Up to 12 months
  Only subjects who are stable for discharge from ICU and have at least 48 consecutive hours of discharge
Number of subjects discharged from ICU | Day 29
  Only subjects who are stable for discharge from ICU and have at least 48 consecutive hours of discharge
ICU/Respiratory Care Center (RCC) free hours | Day 1 to 29
  Only subjects who are stable for discharge from ICU/RCC and have at least 48 consecutive hours of discharge
Changes in Sequential Organ Failure Assessment (SOFA) score from baseline | Baseline, Day 4, 6, 8, 15, 29
  The SOFA is a simple and objective score to evaluate the status of organ dysfunction of six organ systems (respiratory, coagulatory, liver, cardiovascular, renal, and neurologic). A subject is defined as free of organ failure when the SOFA score is zero. The total score of SOFA is 24.
Cumulative vasopressor free days | Day 1 to 29
  The cumulative vasopressor free days are the sum of the days without taking vasopressor up to Day 29 or death.
Cumulative oxygen support free hours | Day 1 to 29
  The cumulative oxygen support free hours are the sum of hours without oxgen support up to Day 29 or death
The net change in c-reactive protein (CRP) from baseline | Baseline, Day 4, 6, 8, 15, and 29
  C-reactive protein is an inflammatory marker
The net change in D-dimer from baseline | Baseline, Day 4, 6, 8, 15, and 29
  D-dimer is an inflammatory marker
The net change in Lactate Dehydrogenase (LDH) from baseline | Baseline, Day 4, 6, 8, 15, and 29
  LDH is an inflammatory marker
The domain scores and total score of 12-item Short Form Survey (SF-12) Quality of Life (QoL) health survey questionnaire | Month 3, 6, 9, 12
  The SF-12 QoL is a self-evaluated measurement of health status. It consists of eight domains and the score of each domain is transformed to a scale from 0 to 100. Zero indicates the worst health status, while 100 indicates the best health status.
Number of subjects who experienced Dose Limiting Toxicity (DLT) | Day 1 to 29
  A DLT is defined as any SAE OR any equal or greater than Grade 3 (CTCAE v5.0) AE judged as MatriPlax-related during Day 1 to 29. The CTCAE (Common Terminology Criteria for Adverse Events) is a classification system used to grade AE.
Incidence of TEAEs (treatment-emergent AEs) and SAEs | 12 months
  The number of TEAEs (treatment-emergent AEs) and SAEs that occur in the study
Number of participants with abnormalities in vital signs | Baseline, Day 1, 4, 6, 8, 15, 29, Month 3, 6, 9, 12
  The vital signs include blood pressure, respiratory rate, oxygen saturation, pulse rate, and body temperature
Number of participants with abnormalities in physical examination | Baseline, Day 1, 4, 6, 8, 15, 29, Month 3, 6, 9, 12
  A physical examination includes general appearance, skin, eyes, ears, nose, throat, head and neck (including thyroid), heart, chest and lungs, abdomen, extremities, lymph nodes, musculoskeletal, neurological system, and other body systems if applicable.
Number of participants with abnormalities in laboratory examination parameters | Baseline, Day 1, 4, 6, 8, 15, 29
  The laboratory examination parameters include hematology (hemoglobin, hematocrit, red blood cell (RBC), platelet, white blood cell (WBC), neutrophils, lymphocytes, monocytes, eosinophils, basophils) and biochemistry (blood urea nitrogen (BUN), creatinine, albumin, total protein, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, C-reactive protein (CRP), prothrombin time (PT), D-dimer, Lactate Dehydrogenase (LDH))
Number of participants with abnormalities in ECG parameters | Baseline, Day 29
  The ECG parameters include ventricular rate, PR interval, QRS interval, and QT interval. Each parameters will be evaluated by the investigator as "Normal", "Abnormal, non-clinical significant (NCS)" or "Abnormal, clinical significant (CS)".

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen MC, Lai KS, Chien KL, Teng ST, Lin YR, Chao W, Lee MJ, Wei PL, Huang YH, Kuo HP, Weng CM, Chou CL. pcMSC Modulates Immune Dysregulation in Patients With COVID-19-Induced Refractory Acute Lung Injury. Front Immunol. 2022 Apr 29;13:871828. doi: 10.3389/fimmu.2022.871828. eCollection 2022. PMID 35585988